CLINICAL TRIAL: NCT01224600
Title: EValuation of Systemic Atherothrombosis in Patients With ARTerial Disease of the Lower Limbs
Acronym: EVART
Status: Completed | Type: Observational
Sponsor: Institut de l'Atherothrombose (Other)
Responsible Party: Sponsor
Other Study IDs: DCIC 0704
Record Dates: First submitted 2010-09-15; First posted 2010-10-20 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral Arterial Disease; Carotid Stenosis; Abdominal Aortic Aneurysm
Keywords: lower limbs; Arterial Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Carotid Stenosis; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: patient with newly diagnosed PAD (< 1 year)
  Interventions: Other: patients with newly diagnosed PAD (<1year)

INTERVENTIONS:
Other: patients with newly diagnosed PAD (<1year) — patients with newly diagnosed PAD (<1year) symptomatic or asymptomatic, without any history of previous coronary nor cerebrovascular event, and with no previous investigation of the aorta and cervical arteries were eligible
  Other Names: arterial disease of the lower limbs; carotid stenosis; aortic aneurysm

SUMMARY:
The purpose of this study is to determine the prevalence and risk factors, at the time of the diagnosis of PAD, for asymptomatic carotid stenosis and abdominal aortic aneurysm.

DETAILED DESCRIPTION:
The EVART study is a prospective epidemiological multicenter cohort study, including patients with newly diagnosed PAD (< 1 year). Initial data on medical history, caracterisation of the PAD (risk factors, main sites and severity of the atherosclerotic lesions),clinical evaluation of undetected previous CV events, standardized US duplex examination of the abdominal aorta and carotid arteries and treatment (type and duration) are collected by the physician into an electronic medical record. A phone follow up at 3 months, 1, 2 and 3 years is realised by the Centre for Clinical Research of Grenoble. Data on mortality, revascularization, treatments prescribed (type and duration), cancer onset, cardiovascular events, carotid stenosis, abdominal aortic aneurysm are collected. All these serious adverse events are documented and reviewed by an independent critical events committee.

ELIGIBILITY:
Inclusion Criteria:

* patient with newly diagnosed PAD < 1 year
* symptomatic or asymptomatic : ABI<0.9 at rest, claudicants with ABI<0.85 after treadmill test, or symptomatic patients (Edimburgh questionnaire or trophic changes) with ABI>1.30

Exclusion Criteria:

* history of previous coronory or cerebrovascular event
* previous investigation of the aorta and cervical arteries
* prisoners
* subjets with no affiliation to the social security system or equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed PAD < 1 year symptomatic or asymptomatic without any hystory of previous coronary nor cerebrovascular event
Sampling Method: Non-Probability Sample
Enrollment: 1056 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
prevalence and risk factors, at the time of the diagnosis PAD, for asymptomatic carotid stenosis and abdominal aortic aneurysm | evaluation during inclusion visit

SECONDARY OUTCOMES:
clinical forms of aortic aneurysm and carotid stenosis, clinical stage of PAD, ABI level, proximal predominance, age, gender, cardiovascular risk factors will be tested like potential aneurysm or carotid stenosis risk factor | evaluation during inclusion visit
frequency of prescription of cardiac consultation,coronarography, stress ECG, stress echo, thallium scan and renal and digestive doppler ultrasound. Frequency of coronary and renal revascularization | evaluation during inclusion visit
frequency of drug prescription (beta blocker, statin,antiplatelet,ICE, other hypolipidaemic...) Non-drug prescription : dietetic, tabagism, rehabilitation for walking and structured therapeutic education, dietary management | evaluation during inclusion visit
incidence and cardiovascular risk factor | 3 months, 1, 2 and 3 years
incidence of thromboembolic disease (symptomatic DVT and/or PE) proved by additional examinations | 3 Months, 1, 2 and 3 years
useful of the screening | 3 years
  decision analysis

CONTACTS AND LOCATIONS:
Overall Officials: Patrick CARPENTIER, Professor, Principal Investigator — University Hospital, Grenoble
Locations (115):
- University hospital Liège, Chênée, Belgium
- France (114):
  - Hospital, Abbeville
  - Office-based Specialist in vascular medecine, Alençon
  - Office-based Specialist in vascular medecine, Ambarès-et-Lagrave
  - University Hospital Amiens, Amiens
  - Office-based Specialist in vascular medecine, Amiens
  - Office-based Specialist in vascular medecine, Annecy
  - Hospital center Armentières, Armentières
  - Office-based Specialist in vascular medecine, Arpajon
  - Office-based Specialist in vascular medecine, Auxerre
  - Office-based Specialist in vascular medecine, Basse-terre (Guadeloupe)
  - Office-based Specialist in vascular medecine, Beauvais
  - Office-based Specialist in vascular medecine, Blagnac
  - Hospital Saint-André, Bordeaux
  - Office-based Specialist in vascular medecine, Bordeaux
  - Hospital center, Boulogne-sur-Mer
  - Office-based Specialist in vascular medecine, Bourg-en-Bresse
  - Office-based Specialist in vascular medecine, Bourgoin
  - Office-based Specialist in vascular medecine, Brest
  - University Hospital Brest, Brest
  - Office-based Specialist in vascular medecine, Bretigny
  - Hospital center, Brive-la-Gaillarde
  - University Hospital Caen, Caen
  - Office-based Specialist in vascular medecine, Cannes
  - Office-based Specialist in vascular medecine, Carcassonne
  - Hospital Antoine Gayraud, Carcassonne
  - Office-based Specialist in vascular medecine, Castres
  - Office-based Specialist in vascular medecine, Ceyrat
  - Office-based Specialist in vascular medecine, Chalon-sur-Saône
  - Office-based Specialist in vascular medecine, Chambéry
  - Office-based Specialist in vascular medecine, Chartres
  - Hospital Center Versailles, Chesnay
  - Office-based Specialist in vascular medecine, Cholet
  - Office-based Specialist in vascular medecine, Clermont-Ferrand
  - Office-based Specialist in vascular medecine, Cluses
  - Office-based Specialist in vascular medecine, Cognac
  - Hospital Center Compiègne, Compiègne
  - Office-based Specialist in vascular medecine, Crolles
  - Office-based Specialist in vascular medecine, Denain
  - Bocage Hospital, Dijon
  - Office-based Specialist in vascular medecine, Ermont
  - Office-based Specialist in vascular medecine, Eu
  - Office-based Specialist in vascular medecine, Fécamp
  - Hospital center Val d'Ariège, Foix
  - Office-based Specialist in vascular medecine, Fort de France
  - Office-based Specialist in vascular medecine, Grenoble
  - University Hospital Grenoble, Grenoble
  - Office-based Specialist in vascular medecine, Issy-les-Moulineaux
  - Office-based Specialist in vascular medecine, La Membrolle-sur-Choisille
  - Office-based Specialist in vascular medecine, La Rochelle
  - Hospital Center Lens, Lens
  - Office-based Specialist in vascular medecine, Levallois-Perret
  - University Hospital Lille, Lille
  - University Hospital Limoges, Limoges
  - Office-based Specialist in vascular medecine, Limoges
  - Office-based Specialist in vascular medecine, Lomme
  - Hospital Saint Philibert, Lomme
  - Office-based Specialist in vascular medecine, Longwy
  - Edouard Herriot Hospital, Lyon
  - Office-based Specialist in vascular medecine, Lyon
  - Office-based Specialist in vascular medecine, Malemort-sur-Corrèze
  - Office-based Specialist in vascular medecine, Maubeuge
  - Hospital of Belfort, Montbéliard
  - Office-based Specialist in vascular medecine, Montélimar
  - Office-based Specialist in vascular medecine, Montluçon
  - University hospital Montpellier, Montpellier
  - Office-based Specialist in vascular medecine, Mulhouse
  - Office-based Specialist in vascular medecine, Nice
  - Office-based Specialist in vascular medecine, Niort
  - Office-based Specialist in vascular medecine, Noumea
  - Hospital Center, Orléans
  - Office-based Specialist in vascular medecine, Orléans
  - Hospital center Territorial Mamao, Papeete
  - Office-based Specialist in vascular medecine, Paris
  - Office-based Specialist in vascular medecine, Perpignan
  - Hospital Center, Périgueux
  - Office-based Specialist in vascular medecine, Péronne
  - Office-based Specialist in vascular medecine, Pontcharra
  - Office-based Specialist in vascular medecine, Pornic
  - Office-based Specialist in vascular medecine, Puilboreau
  - Office-based Specialist in vascular medecine, Rambouillet
  - Office-based Specialist in vascular medecine, Rochefort
  - Office-based Specialist in vascular medecine, Rodez
  - Hospital center Rodez, Rodez
  - Office-based Specialist in vascular medecine, Rouen
  - Office-based Specialist in vascular medecine, Saint-Aubin-de-Médoc
  - Office-based Specialist in vascular medecine, Saint-Aubin-sur-Scie
  - Office-based Specialist in vascular medecine, Saint-Benoît
  - Office-based Specialist in vascular medecine, Saint-Etienne
  - University Hospital Saint Etienne, Saint-Etienne
  - Memorial Hospital, Saint-Lô
  - Office-based Specialist in vascular medecine, Saint-Lô
  - Office-based Specialist in vascular medecine, Saint-Priest
  - Hospital, Saint-Quentin
  - Office-based Specialist in vascular medecine, Sallanches
  - Office-based Specialist in vascular medecine, Sarcelles
  - Office-based Specialist in vascular medecine, Sarrebourg
  - Office-based Specialist in vascular medecine, Sarreguemines
  - Office-based Specialist in vascular medecine, Savigny-sur-Orge
  - Office-based Specialist in vascular medecine, Sélestat
  - Office-based Specialist in vascular medecine, Strasbourg
  - Office-based Specialist in vascular medecine, Toulon
  - University Hospital Rangueil, Toulouse
  - Office-based Specialist in vascular medecine, Toulouse
  - Office-based Specialist in vascular medecine, Tours
  - Office-based Specialist in vascular medecine, Trélazé
  - Office-based Specialist in vascular medecine, Trois-Rivières (Guadeloupe)
  - Office-based Specialist in vascular medecine, Vannes
  - Office-based Specialist in vascular medecine, Versailles
  - Office-based Specialist in vascular medecine, Vienne
  - Office-based Specialist in vascular medecine, Villeurbanne
  - Office-based Specialist in vascular medecine, Vincennes
  - Office-based Specialist in vascular medecine, Vizille
  - Office-based Specialist in vascular medecine, Voiron
  - Office-based Specialist in vascular medecine, Wissembourg